CLINICAL TRIAL: NCT00854178
Title: Toxicogenomic and Immunocytotoxic Effects of Propofol and Isoflurane Anesthetics in Patients Undergoing Elective Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Mariana Gobbo Braz, São Paulo State University, UNESP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: upeclin/HC/FMB-Unesp-20
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Patients in Good Health; Types of General Anesthesia; DNA Damage
Keywords: isoflurane; propofol; genotoxicity; gene expression; cytokines; apoptosis
MeSH Terms: interventions — Propofol; Isoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental)
  Interventions: Drug: Comparison of two anesthetic drugs

INTERVENTIONS:
Drug: Comparison of two anesthetic drugs — Isoflurane 1,0 minimum alveolar concentration Propofol 2mg/kg and 4ug/ml
  Other Names: Diprivan; Isoflurane

SUMMARY:
The purpose of this study is to evaluate if the anesthetics propofol and isoflurane can damage DNA, induce apoptosis, change expression of genes related to apoptosis and DNA repair and change cytokines profile in patients submitted to elective surgery.

DETAILED DESCRIPTION:
It is expected that the results provide relevant information to understand the possible adverse effects of anesthetics and contribute to the establishment of strategies aimed at reducing the risks to exposed individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients in good health American Society of Anesthesia status physical I
* elective minor surgery
* general anesthesia

Exclusion Criteria:

* smokers
* alcoholics
* previous medication or radiation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of genotoxicity, gene expression, apoptosis and cytokines profile | within 1 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mariana G Braz, MsC, Principal Investigator — Department of Pathology, Botucatu Medical School, São Paulo State University, UNESP
Locations (1):
- Botucatu Medical School, UNESP, Botucatu, São Paulo, Brazil